CLINICAL TRIAL: NCT02905487
Title: Relation Entre diabète Gestationnel et Adipocytokines Inflammatoires Chez Des mères obèses et Leur Nouveau-né à l'Accouchement
Brief Title: Relationship Between Gestational Diabetes Mellitus and Inflammatory Adipocytokins in Obese Mothers and Their Newborn at Delivery
Acronym: ADIPOGEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/CHU/ADIPOGEST
Record Dates: First submitted 2016-09-12; First posted 2016-09-19 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes, Gestational
Keywords: Gestational Diabetes Mellitus; Obesity; Adipocytokin
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Leptin, adiponeptin, TNF-alpha, Interleukin-6, CRP and C-peptide blood levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GDM: Mother-child pairs from mothers with GDM diagnosis (ADA, 2012)
- No GDM: Mother-child pairs from mothers without GDM diagnosis (ADA, 2012)

SUMMARY:
ADIPOGEST study aims at comparing circulating levels of inflammatory adipocytokins and C-reactive protein in obese women and their newborn at delivery whether exposed or not to Gestational Diabetes Mellitus (GDM)

DETAILED DESCRIPTION:
ADIPOGEST is a cross sectional study in which mothers are divided into 2 groups : exposed and unexposed to GDM, matched on pregestational BMI, date of delivery and child gender.

Mothers are recruited in the maternity ward of the University Hospital in South of Reunion Island.

It is planned a conveniance sample of 20 mother-child pairs per group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Obese women (BMI : 30 kg/m² or more)
* Aged over 18 years
* With single pregnancy
* With alive newborn at 37 weeks of amenorrhea or more
* With informed consent

Exclusion Criteria:

* Smoker
* Treatments by corticoïds or thyroid hormons
* Overt diabetes
* Complicated pregnancy
* Premature delivery threat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mother-child pairs from obese women with GDM or not
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Blood levels of leptin in mother and her child | 2 years
Blood levels of adiponectin in mother and her child | 2 years
Blood levels of IL-6 in mother and her child | 2 years
Blood levels of TNF-alpha in mother and her child | 2 years
Blood levels of C- Reactive Protein in mother and her child | 2 years

SECONDARY OUTCOMES:
Blood level of C-peptide in mother | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Universitaire de La Réunion, Saint-Pierre, France